CLINICAL TRIAL: NCT01362907
Title: Clinical Comparison of Silicone Hydrogel and HEMA-based Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-347-C-013
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Results first posted 2012-08-03 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delefilcon A / etafilcon A (Other): Delefilcon A contact lenses worn first, with etafilcon A contact lenses worn second. Both products worn bilaterally on a daily wear, daily disposable basis for one week each.
  Interventions: Device: Delefilcon A contact lens; Device: Etafilcon A contact lens
- Etafilcon A / delefilcon A (Other): Etafilcon A contact lenses worn first, with delefilcon A contact lenses worn second. Both products worn bilaterally on a daily wear, daily disposable basis for one week each.
  Interventions: Device: Delefilcon A contact lens; Device: Etafilcon A contact lens

INTERVENTIONS:
Device: Delefilcon A contact lens — Investigational, silicone hydrogel, single vision, soft contact lens for daily disposable wear
  Other Names: DAILIES® Total1®
Device: Etafilcon A contact lens — Commercially marketed, HEMA-based, single vision, soft contact lens for daily disposable wear
  Other Names: 1-DAY ACUVUE® MOIST™

SUMMARY:
The purpose of this trial was to compare the performance of an investigational daily disposable contact lens to a commercially available daily disposable contact lens.

ELIGIBILITY:
Inclusion Criteria:

* Normal eyes with no use of ocular medications.
* Be of legal age of consent and sign Informed Consent document. If under legal age of consent, legally authorized representative must sign Informed Consent document and subject must sign Assent document.
* Willing and able to wear spherical contact lenses for protocol-specified timeframe within the available range of powers (-1.00 D to -6.00D in 0.25D steps).
* Visual acuity with study lenses 20/25 or better.
* Cylinder less than or equal to 0.75 D.
* Currently wearing daily disposable lenses.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Anterior segment infection, inflammation, or abnormality.
* Any active anterior segment ocular disease that would contraindicate contact lens wear.
* Any use of systemic medications for which contact lens wear could be contraindicated as determined by the investigator.
* History of refractive surgery or irregular cornea.
* Eye injury within twelve weeks immediately prior to enrollment for this trial.
* Currently enrolled in any clinical trial.
* Other protocol-defined exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 4 US private practices.
Period: Period 1, One Week
Arm/Group | Delefilcon A / Etafilcon A | Etafilcon A / Delefilcon A
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Period 2, One Week
Arm/Group | Delefilcon A / Etafilcon A | Etafilcon A / Delefilcon A
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: All enrolled participants
Arm/Group | Overall
Number analyzed (Participants) | 40
Age Continuous [Mean (Standard Deviation); unit: years] | 32.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Corrected Distance Monocular Visual Measurement Reported as Visual Acuity (VA)
Description: As tested for each eye individually while wearing study lenses. VA was measured using a Snellen chart, which was converted into logMAR units (logarithm of the minimum angle of resolution). A 20/20 Snellen acuity equated to a logMAR acuity of 0.0 and was considered normal distance eyesight. Positive logMAR values indicated poorer vision, and negative values denoted better visual acuity.
Time Frame: 1 week of wear, replacing lenses daily
Population: All enrolled and dispensed participants.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- Delefilcon A: Delefilcon A contact lenses worn bilaterally on a daily wear, daily disposable basis for one week.
- Etafilcon A: Etafilcon A contact lenses worn bilaterally on a daily wear, daily disposable basis for one week.
Arm/Group | Delefilcon A | Etafilcon A
Number analyzed (Participants) | 40 | 40
Number analyzed (eyes) | 80 | 80
logMAR | -0.02 (0.06) | -0.02 (0.05)

2. Primary Outcome: Overall Comfort
Description: As interpreted by the participant and recorded on a questionnaire as a single, retrospective evaluation of 1 week of wear time. Overall comfort was evaluated binocularly and rated on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 1 week of wear, replacing lenses daily
Population: All enrolled and dispensed participants.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Etafilcon A
Number analyzed (Participants) | 40 | 40
Units on a scale | 9.0 (1.5) | 8.1 (1.6)

3. Primary Outcome: Overall Vision Quality
Description: As interpreted by the participant and recorded on a questionnaire as a single, retrospective evaluation of 1 week of wear time. Overall vision quality was evaluated binocularly and rated on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 1 week of wear, replacing lenses daily
Population: All enrolled and dispensed participants.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Etafilcon A
Number analyzed (Participants) | 40 | 40
Units on a scale | 9.4 (1.0) | 8.9 (1.2)

4. Primary Outcome: Overall Handling
Description: As interpreted by the participant and recorded on a questionnaire as a single, retrospective evaluation of 1 week of wear time. Overall handling was evaluated binocularly and rated on a 10-point scale, with 1 being difficult and 10 being easy.
Time Frame: 1 week of wear, replacing lenses daily
Population: All enrolled and dispensed participants.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Etafilcon A
Number analyzed (Participants) | 40 | 40
Units on a scale | 8.5 (1.9) | 8.6 (1.4)

5. Secondary Outcome: Overall Lens Fit
Description: As assessed for each eye individually by the investigator using a biomicroscope, which magnifies the appearance of the contact lens on the participant's eye. Lens fit is reported on a 5-point scale, with 2=unacceptably loose, 1=acceptably loose, 0=optimal, -1=acceptably tight, and -2=unacceptably tight.
Time Frame: 1 week of wear, replacing lenses daily
Population: All enrolled and dispensed participants.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | Delefilcon A | Etafilcon A
Number analyzed (Participants) | 40 | 40
Number analyzed (eyes) | 80 | 80
Units on a scale | -0.1 (0.5) | 0.1 (0.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the trial: 1 month.
Description: The safely population included all enrolled and exposed participants.
Arm/Group | Delefilcon A | Etafilcon A
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.